CLINICAL TRIAL: NCT07194291
Title: Menstrual Cycle Changes in Adolescent Girls With Diabetes
Brief Title: Menses&Change in Diabetic Girl
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Zeinab Megahed Mohammed Shelgamy, Principal Investigator, Assiut University
Other Study IDs: Menses&Change in diabetic Girl
Record Dates: First submitted 2025-09-03; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Adolescent Girls; Diabete Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Follow up of female sexual function — We follow up menstrual changes in diabetic adolescent girls to improve the outcome

SUMMARY:
To assess menstraul cycle changes in adolescent girls with diabetes and to find out the various risk factors

DETAILED DESCRIPTION:
Type 1 diabetes mellitus (T1DM) is the result of autoimmunity mediated destruction of pancreatic beta cells, ultimately causing insulin deficiency and, consequently, hyperglycemia .

Typically the diagnosis of T1DM is made in childhood or adolescence,but about 40% of affected individuals are diagnosed in adulthood.

Hyperglycemia-related complications can contribute to impairment of endocrine axes, such as the hypothalamic pituitary gonadal (HPG) axis .

Historically, before the introduction of insulin replacement therapy, prepubertal girls wh developed T1DM rarely showed normal sexual development, exhibiting primary amenorrhea .

Although the introduction of insulin drastically changed the natural history of T1DM, allowing restoration of the HPG physiology, menarche delay remained as a typical sign in girls with T1DM .

In addition, women with T1DM report a higher incidence of menstrual irregularities >30%

compared with control subjects without diabetes .

Accordingly, signs and symptoms of androgen excess, such as acne and hirsutism, are more frequent in women with T1DM than in their age-matched counterparts

These interconnected abnormalities contribute to the reduced fertility observed in women with T1DM, as characterized by fewer pregnancies and live births and earlier menopause compared with women without diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Girls with diabetes diagnosed based on ADA guidelines Who reatched menarche of at least 1year duration [14]]
2. Another comparable number of age matched non_diabetic girls will be included as controls.

3/Female adolescents aged 10-18 years

Exclusion Criteria:

1. Girls Known thyroid disease or other endocrine disorders affecting menstruation
2. Girls taking medications that may affect menstrual cycles like Use of hormonal therapy (e.g., oral contraceptive pills) within the last 6 months
3. Menstraul irregularitis prior to diagnosis of diabetes

Ages: 10 Years to 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Study Population: Adolescent girls with diabetes are at higher risk of menstrual cycle irregularities due to metabolic, hormonal, and nutritional factors. Early recognition of these changes is essential to improve reproductive health and overall quality of life.
Sampling Method: Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with menstrual irregularities | 12 months (from enrollment)
  Menstrual cycle characteristics (cycle length, frequency, and regularity) will be documented using a structured menstrual diary and standardized questionnaire. Menstrual irregularity will be defined as the presence of oligomenorrhea (cycle length > 35 days), amenorrhea (≥ 3 months without menstruation), or polymenorrhea (cycle length < 21 days). Data will be summarized as the number and percentage of participants meeting any of these criteria.

SECONDARY OUTCOMES:
Association of menstrual irregularities with HbA1c and BMI | 12 months (from enrollment)
  HbA1c levels and body mass index (BMI) will be recorded at baseline and at 12 months. Data will be analyzed to assess correlations between menstrual irregularities and glycemic control (HbA1c, %) and nutritional status (BMI, kg/m²).

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ghitha N, Vathania N, Wiyono L, Pulungan A. Delayed menarche in children and adolescents with type 1 diabetes mellitus: a systematic review and meta-analysis. Clin Pediatr Endocrinol. 2024;33(3):104-112. doi: 10.1297/cpe.2023-0058. Epub 2024 Apr 19. PMID 38993726
- [Background] Whitworth KW, Baird DD, Stene LC, Skjaerven R, Longnecker MP. Fecundability among women with type 1 and type 2 diabetes in the Norwegian Mother and Child Cohort Study. Diabetologia. 2011 Mar;54(3):516-22. doi: 10.1007/s00125-010-2003-6. Epub 2010 Dec 19. PMID 21170514
- [Background] Gu YH, Yokoyama K, Mizuta K, Tsuchioka T, Kudo T, Sasaki H, Nio M, Tang J, Ohkubo T, Matsui A. Stool color card screening for early detection of biliary atresia and long-term native liver survival: a 19-year cohort study in Japan. J Pediatr. 2015 Apr;166(4):897-902.e1. doi: 10.1016/j.jpeds.2014.12.063. Epub 2015 Feb 11. PMID 25681196
- [Background] Samara-Boustani D, Colmenares A, Elie C, Dabbas M, Beltrand J, Caron V, Ricour C, Jacquin P, Tubiana-Rufi N, Levy-Marchal C, Delcroix C, Martin D, Benadjaoud L, Jacqz Aigrain E, Trivin C, Laborde K, Thibaud E, Robert JJ, Polak M. High prevalence of hirsutism and menstrual disorders in obese adolescent girls and adolescent girls with type 1 diabetes mellitus despite different hormonal profiles. Eur J Endocrinol. 2012 Feb;166(2):307-16. doi: 10.1530/EJE-11-0670. Epub 2011 Nov 29. PMID 22127492
- [Background] Codner E, Soto N, Merino PM. Contraception, and pregnancy in adolescents with type 1 diabetes: a review. Pediatr Diabetes. 2012 Feb;13(1):108-23. doi: 10.1111/j.1399-5448.2011.00825.x. Epub 2011 Oct 13. PMID 21995767
- [Background] Strotmeyer ES, Steenkiste AR, Foley TP Jr, Berga SL, Dorman JS. Menstrual cycle differences between women with type 1 diabetes and women without diabetes. Diabetes Care. 2003 Apr;26(4):1016-21. doi: 10.2337/diacare.26.4.1016. PMID 12663566
- [Background] Kjaer K, Hagen C, Sando SH, Eshoj O. Epidemiology of menarche and menstrual disturbances in an unselected group of women with insulin-dependent diabetes mellitus compared to controls. J Clin Endocrinol Metab. 1992 Aug;75(2):524-9. doi: 10.1210/jcem.75.2.1639955.
- [Background] Green A, Hauge M, Holm NV, Rasch LL. Epidemiological studies of diabetes mellitus in Denmark. II. A prevalence study based on insulin prescriptions. Diabetologia. 1981 Apr;20(4):468-70. doi: 10.1007/BF00253409. PMID 7016641
- [Background] Trzeciak B. [Effect of diabetes mellitus on the incidence of abnormal genital bleedings in women]. Ginekol Pol. 1978 Feb;49(2):119-23. No abstract available. Polish. PMID 648900
- [Background] Yeshaya A, Orvieto R, Dicker D, Karp M, Ben-Rafael Z. Menstrual characteristics of women suffering from insulin-dependent diabetes mellitus. Int J Fertil Menopausal Stud. 1995 Sep-Oct;40(5):269-73. PMID 8556032
- [Background] BERGQVIST N. The gonadal function in female diabetics. Acta Endocrinol Suppl (Copenh). 1954;19:1-20. No abstract available. PMID 13147722
- [Background] Arrais RF, Dib SA. The hypothalamus-pituitary-ovary axis and type 1 diabetes mellitus: a mini review. Hum Reprod. 2006 Feb;21(2):327-37. doi: 10.1093/humrep/dei353. Epub 2005 Oct 20. PMID 16239312
- [Background] American Diabetes Association. 2. Classification and Diagnosis of Diabetes: Standards of Medical Care in Diabetes-2021. Diabetes Care. 2021 Jan;44(Suppl 1):S15-S33. doi: 10.2337/dc21-S002. PMID 33298413
- [Background] Richardson SJ, Pugliese A. 100 YEARS OF INSULIN: Pancreas pathology in type 1 diabetes: an evolving story. J Endocrinol. 2021 Dec 9;252(2):R41-R57. doi: 10.1530/JOE-21-0358. PMID 34755679
- [Background] Paschou SA, Papadopoulou-Marketou N, Chrousos GP, Kanaka-Gantenbein C. On type 1 diabetes mellitus pathogenesis. Endocr Connect. 2018 Jan;7(1):R38-R46. doi: 10.1530/EC-17-0347. Epub 2017 Nov 30. PMID 29191919